CLINICAL TRIAL: NCT04145544
Title: A Prospective, Randomized, Controlled Multi-center Study of ArtiFascia® Dural Repair Patch Compared With Commercially Available Dural Substitutes- NEOART Study.
Brief Title: A Prospective, Randomized, Controlled Multi-center Study of ArtiFascia® Dural Repair Patch Compared With Commercially Available Dural Substitutes. To Evaluate the Safety and Effectiveness of ArtiFascia® in Subjects Requiring Dural Repair.
Acronym: NEOART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurami Medical Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARTIFASCIA® DURAL REPAIR PATCH
Record Dates: First submitted 2019-10-21; First posted 2019-10-30 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dural Tear; Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Procedure was performed under general anesthesia. The subjects underwent the planned surgery. At the end of the surgery, the investigator used the ArtiFascia® patch. Implantation of the ArtiFascia® was according to clinical discretion of the physician, and in compliance with ArtiFascia® instructions for use.
  Post operation the subject stayed at the hospital according to site standards and physician discretion.
  Interventions: Device: Implantation of the ArtiFascia®
- Control (Active Comparator): Same procedure as for the treatment arm but using a commercial suturable dural substitute.
  Implantation of the commercial suturable dural substitute was according to clinical discretion of the physician, and in compliance with each specific device instructions for use.
  Interventions: Device: Implantation of other commercial suturable dural substitute

INTERVENTIONS:
Device: Implantation of the ArtiFascia® — Following are the general instructions for use for the ArtiFascia®:
  * Cut the ArtiFascia® to the required shape under aseptic conditions
  * Apply ArtiFascia® to the damaged area
  * Suture the ArtiFascia® in place
  * Suture bites should be taken 2-3 millimeters from the edges of the implant. Either a running suture or interrupted stitches' technique may be used, depending on clinical conditions or surgeon's decision.
  Important Note: If clinically possible, do not use dural adhesive or sealants as it is an uncontrolled variable, that can influence the results.
  Arms: Treatment arm
Device: Implantation of other commercial suturable dural substitute — Implantation of the commercial suturable dural substitute will be according to clinical discretion of the physician, and in compliance with each specific device instructions for use. Detailed instructions are in the instructions for use
  Arms: Control

SUMMARY:
The objective of this study was to evaluate the safety and effectiveness of ArtiFascia® in comparison with commercially available dural substitutes in subjects requiring Dural repair following neurosurgery.

Subjects with planned cranial neurosurgery participated in this study. During the surgery the dura is likely to be cut and damaged. A damaged dura can cause a leakage of brain fluids (cerebrospinal fluid [CSF] leakage) and increase the risk of infections. The damaged dura can be fixed with dural patch like ArtiFascia®. ArtiFascia® is a bioabsorbable medical synthetic dural replacement that aids in the regeneration of a new dura. Furthermore, it incorporates a sealing layer capable of minimizing CSF leakage and infection.

DETAILED DESCRIPTION:
A Prospective, randomized, controlled multi-center study of ArtiFascia® Dural repair patch compared with commercially available dural substitutes- NEOART Study.

The dura mater is a fibrous connective tissue that surrounds the nervous system (brain and spinal cord) and provides a mechanical barrier that contains the cerebrospinal fluid (CSF). The dura mater may be damaged as a result of trauma or planned surgery. When dural defects cannot be repaired by primary closure, a dural substitute must be utilized in order to reduce CSF leakage.

There are devices that have been used as dural substitutes. Among the devices that are based on natural raw materials, collagen-based matrices are widely used. Although collagen was proven to be biocompatible, using collagen-based materials still possess several limitations such as CSF leaks. Synthetic dural substitutes are also used to repair dura mater. The most widely used raw-material for these synthetic products are polyesters - resorbable and biocompatible polymers. There are several dural substitutes based on synthetic polyesters that were successfully tested pre-clinically as well as in human studies.

Sponsor of this study has developed the ArtiFascia®. ArtiFascia® is a polymeric synthetic dural substitute that is absorbed by the body.

Before the study, all subjects underwent neurological assessment. Only subjects that were found to be suitable to participate in the study, and agree to participate, were randomly allocated into one of the following groups:

* Experimental group (ArtiFascia® device);
* Control group (Other commercially available suturable dural substitutes).

The Sponsor was blinded to treatment. The subjects underwent the planned surgery and at the end the investigator used ArtiFascia® patch or standard dural substitute to repair the damaged Dura. ArtiFascia® graft was placed in areas where the native dural layer was damaged or missing. ArtiFascia® was applied via a routine and well-known procedure, using a suturing technique. After implantation, the porous fibrous structure of ArtiFascia® provides a scaffold, which enables infiltration of fibroblasts and cells from the intact tissue, ultimately replacing damaged dural tissue. The patch is expected to resorb within a few months and to be replaced by the native tissue with complete dural closure.

During the surgery and until subject's release from the hospital the subject's health was closely monitored. Before the discharge subjects underwent neurological examination. Subjects had been followed up at 4-6 weeks and at 6 months post surgery.

At each follow up visit physical and neurological examinations were performed. Radiographic Evaluation (Magnetic Resonance Imaging) was performed at 6 months post operation.

A total of 92 subjects from 7 sites in Europe were enrolled and implanted with test or control device.

The primary endpoint was achieved when the final study subject has completed a 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject between the ages of 18-75
2. Subject is scheduled for an elective cranial surgery with a dural damage that can be completely repaired/closed by a suture-able dural substitute (ArtiFascia device or other commercially available dural substitutes)
3. Subject has undergone radiographic imaging (such as, MRI) in the past 6 months before enrolment
4. Surgical wound is expected to be Class I/clean
5. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
6. Subject is able and willing to adhere to the required follow-up visits and testing

Exclusion Criteria:

1. Pregnant women or interest in becoming pregnant during the duration of the study
2. Subject has known hydrocephalus
3. Subject is unable to undergo MRI after the surgery
4. Subject's life expectancy is less than 12 months
5. Subject has a local or systemic infection (e.g. urinary tract infection (UTI), active pneumonia) or evidence of any surgical site infection, fever > 38.3℃, positive blood culture and/or a positive chest x-ray for acute infectious process
6. Subject will require use of dural adhesive or sealant
7. Subject is intended to undergo craniectomy wherein bone flap will not be returned
8. Subject with suspected low success in wound healing due to past treatments (e.g. chemotherapy, radiation therapy, severe diabetes etc.) or other conditions (e.g. severe peripheral vascular disease, long standing steroids treatment)
9. Subject has been clinically diagnosed with malignancy (other than basal cell carcinoma or low-grade glioma), uncontrolled diabetes (A1C>6.5%), sepsis, systemic collagen disease.
10. Subject had chemotherapy and/or radiotherapy in the past 12 weeks before surgery or is planned to have chemotherapy or radiotherapy less than 12 weeks after surgery.
11. Subject is an acute cranial trauma surgical case
12. Subjects with a concurrent disease that would place the patient in excessive risk to the planned surgery
13. Subject had a previous neurosurgery in the same anatomical site
14. Subject with other undesirable symptoms defined by the principal investigator
15. Patient has clinically significant coagulopathy as determined by the surgeon
16. Subject is participating in another clinical trial using similar investigational devices/drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Czechia (2):
  - St. Anne's University Hospital Brno, Brno
  - Neurochirurgická klinika Přednosta FN Olomouc, Olomouc
- Rabin Medical Center (Beilinson, Hasharon), Petah Tikva, Israel
- Poland (2):
  - Medical University of Gdańsk, Gdansk
  - Barlicki University Hospital, Lodz
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical trial was performed in 8 European medical centers (Poland, Czech Republic, Spain and Belgium) and in 1 Israeli medical center. Subjects were enrolled from January 2020 to January 2022.
Pre-assignment Details: A total of 92 subjects met the inclusion/exclusion criteria, were randomized and enrolled. Of those 92 subjects, 89 received surgical treatment. Of those 89 treated subjects, 85 completed the study.
Groups:
- Treatment Arm- ArtiFascia® Patch: The treatment arm consists of subjects who were implanted with ArtiFascia® Dura Replacement device.
- Control-Other Commercial Suturable Dural Substitute: The control arm consists of other commercial suturable dural substitute, including:
  Neuro-patch, ReDura, Tachosil, Tutopatch and Duragen.
Period: Overall Study
Arm/Group | Treatment Arm- ArtiFascia® Patch | Control-Other Commercial Suturable Dural Substitute
Started | 63 | 29
Treated | 62 | 27
Completed | 58 | 27
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: Men and women between the ages of 18-75 scheduled for an elective cranial surgery that requires dural repair, meet all the inclusion and none of the exclusion criteria.
Groups:
- Treatment Arm-ArtiFascia® Graft: The treatment arm consists of patients implanted with ArtiFascia® graft following cranial surgery.
- Control-Other Commercial Suturable Dural Substitute: The control arm consists of patients implanted with other commercial suturable dural substitute, including: Neuro-patch, ReDura, Tachosil, Tutopatch and Duragen.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm-ArtiFascia® Graft | Control-Other Commercial Suturable Dural Substitute | Total
Number analyzed (Participants) | 63 | 29 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 48 | 23 | 71
  >=65 years | 15 | 5 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 21 | 64
  Male | 20 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 4 | 18
  Not Hispanic or Latino | 49 | 25 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 62 | 29 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 3 | 2 | 5
  Czechia | 19 | 9 | 28
  Poland | 28 | 12 | 40
  Spain | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Absence of Cerebrospinal Fluid Fistula (Drainage From Wound or Sinus) and Pseudo-meningocele Within 6 Months Post-operative as Evaluated by MRI Imaging.
Description: The primary end point will be assessed by evaluating the absence of cerebrospinal fluid fistula (drainage from wound or sinus) and pseudo-meningocele post-operative as evaluated by MRI imaging and physical examination of the surgical site.
Time Frame: 6 month.
Measure: Count of Participants; unit: Participants
Groups:
- Control-Other Commercial Suturable Dural Substitute: The control arm consists of subjects implanted with other commercial suturable dural substitute, including: Neuro-patch, ReDura, Tachosil, Tutopatch and Duragen.
- Treatment Arm-ArtiFascia® Graft: The treatment arm consists of subjects implanted with ArtiFascia® graft following cranial surgery.
Arm/Group | Control-Other Commercial Suturable Dural Substitute | Treatment Arm-ArtiFascia® Graft
Number analyzed (Participants) | 27 | 58
Participants
  Presence of cerebrospinal fluid fistula and Pseudomeningocele | 0 | 0
  No events of cerebrospinal fluid fistula and Pseudomeningocele | 27 | 58

2. Secondary Outcome: Wound Healing Assessment
Description: Clean and/or fully healed vs. Infected. Evaluation of wound will be done in physical examination: clean and/or fully healed/ infected. If wound is infected additional assessment of mild/moderate/severe will be done.
Time Frame: 6 month follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Device Handling Characteristics as Reported by a User Experience Questionnaire
Description: The following scoring system was used for the evaluation:
  1) Device ease of use, suturing and cutting were evaluated on a scale of 1=Easy to 5=Difficult. 2) Device strength and seal quality (during implantation) were scored on scale of 1=Low to 5=High.
Time Frame: On the day of the surgical procedure
Reporting Status: Not Posted

4. Secondary Outcome: Radiological Imaging at 6 Months for Additional Findings at Implant Site
Description: The rate of each of the following: Extracerebral fluid accumulation, pseudomeningocele, adhesion formation, brain edema adjacent to device implant site, abnormal thickening at implantation site and new membrane (scar) formation.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm-ArtiFascia® Graft | Control-Other Commercial Suturable Dural Substitute
Number analyzed (Participants) | 58 | 27
Participants
  Present measures | 1 | 3
  No findings presence | 57 | 24

ADVERSE EVENTS:
Time Frame: 2.5 years
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs, including an abnormal laboratory findings in subjects, users or other persons, in the context of a clinical investigation, whether or not related to the investigational device.
Arm/Group | Treatment Arm-ArtiFascia® Graft | Control-Other Commercial Suturable Dural Substitute
All-Cause Mortality (participants affected / at risk) | 1/63 | 0/29
Serious Adverse Events (participants affected / at risk) | 9/63 | 3/29
Other Adverse Events (participants affected / at risk) | 26/63 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm-ArtiFascia® Graft (N=63) | Control-Other Commercial Suturable Dural Substitute (N=29)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) — Postoperative paresis of the right facial nerve. Not related to device, possibly related to procedure.
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — B-cell non-Hodgkin lymphoma. Not related to device nor procedure
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Lambda light chain myeloma. Not related to device nor procedure
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Tumor regrowth in right orbit - possibly a connective tissue disease. Not related to device nor procedure
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) — intracerebral hemorrhage. Not related to device nor procedure
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) — epidural abscess. Not related to device, possibly related to procedure
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Pneumonia. Not related to device nor procedure
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) — Cardiorespiratory arrest. Not related to device nor procedure
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — Seizure. Not related to device, probably related to procedure
Vasospasm (Vascular disorders) | 0 (0) | 1 (1) — Vasospasm. Not related to device, causally related to procedure.
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Diagnosis of cerebral metastasis of renal carcinoma. Not related to device nor procedure.
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) — Hemiplegia - left sided. Not related to device, causally related to procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm-ArtiFascia® Graft (N=63) | Control-Other Commercial Suturable Dural Substitute (N=29)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) — Amnesia of faces. Not related to device nor procedure.
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) — Right ptosis. Not related to device, causally related to procedure.
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1) — Postoperative paresis of the right facial nerve. Not related to device, probably related to procedure.
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) — Taste disturbance, salty aftertaste. Not related to device nor procedure
Skin infection (Infections and infestations) | 1 (1) | 0 (0) — a small puncture infection at the site of one suture, caused by the doctor leaving a fragment of the suture in the skin. The fragment has been removed. The wound heals properly. Not related to device, possibly related to procedure.
Eye swelling (Eye disorders) | 0 (0) | 1 (1) — Swelling of the left eyeball. Not related to device, causally related to procedure.
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) — Paresis of the right facial nerve. Not related to device nor procedure.
Vith nerve paresis (Nervous system disorders) | 1 (1) | 0 (0) — Features of left abducens nerve paresis. Not related to device, probably related to procedure.
Mydriasis (Eye disorders) | 1 (1) | 0 (0) — Left pupil dilatation. Not related to device nor procedure.
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) — Subgaleal collection of cerebrospinal fluid. Probably related to device and procedure.
Inflammation (General disorders) | 0 (0) | 1 (1) — Inflammatory reaction. Not related to device nor procedure.
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hyperglycemia. Not related to device nor procedure
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) — Hypoaesthesia face. Not related to device, possibly related to procedure.
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) — Recurrent sinusitis maxillaris. Not related to device nor procedure.
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Left lower extremity weakness. Not related to device nor procedure.
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Headache. Not related to device nor procedure.
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) — Epileptic fit with post-ictal transient paresis of left lower extremity. Not related to device nor procedure
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) — Mild subgaleal fluid collection - chronic bleeding. Possibly related to device, not related to procedure
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Seizure. Not related to device nor procedure
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) — Hemiparesis progression. Not related to device nor procedure
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hematoma at the incision site. Not related to device, probably related to procedure.
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) — Epileptic fit. Not related to device, possibly related to procedure.
Subgaleal haemorrhage (Vascular disorders) | 1 (1) | 0 (0) — Subgaleal fluid accumulation with external leakage of the fluid - chronic bleeding. Not related to device, causally related to procedure.
Possible dementia Dementia (Nervous system disorders) | 1 (1) | 0 (0) — Possible dementia. Not related to device nor procedure
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Post procedural edema. Not related to procedure nor device.
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1) — Absence seizures. Not related to device nor procedure
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Retroauricular skin lesion 6mm nodular image. Not related to device nor procedure.
Cranial nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) — Paralysis of the VI + V cranial pair. Not related to device nor procedure.
Horner's syndrome (Nervous system disorders) | 1 (1) | 0 (0) — Horner syndrome. Not related to device nor procedure.
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) — Axonopathy of the right trigeminal nerve. Not related to device nor procedure.
Diplopia (Eye disorders) | 1 (1) | 0 (0) — Diplopia. Not related to device nor procedure
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Unknown hypophyseal microincidentaloma. Not related to device nor procedure.
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) — Anxiety-depressive adaptive disorder. Not related to device nor procedure.
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Polyuria Not related to device nor procedure.
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 1 (1) — Right hemianopsia. Not related to device nor procedure.
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) — Respiratory infection. Not related to device nor procedure.
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) — Takotsubo myocardiopathy. Not related to device nor procedure.
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) — Decreased level of consciousness. Not related to device nor procedure.
Epilepsy (Nervous system disorders) | 3 (3) | 0 (0) — Epileptic seizure. Not related to device, causally related to procedure.

LIMITATIONS AND CAVEATS:
No limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04145544/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04145544/SAP_001.pdf